CLINICAL TRIAL: NCT01372917
Title: Evaluating Sterile Human Acellular Dermal Matrix in Immediate Expander-Based Breast Reconstruction: A Multi-centered Prospective Cohort Study
Brief Title: Evaluating AlloMax in Immediate Expander-Based Breast Reconstruction Study
Status: Completed | Type: Observational
Sponsor: National Center for Plastic Surgery, Virginia (Other)
Collaborators: Inova Health Care Services (Other); Ohio State University Comprehensive Cancer Center (Other); Walter Reed Army Medical Center (U.S. Federal Agency); C. R. Bard (Industry)
Responsible Party: Principal Investigator, Mark L. Venturi, MD FACS, Physician, National Center for Plastic Surgery, Virginia
Other Study IDs: 11.064
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Malignant Neoplasm of the Breast; Acquired Absence of the Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A 1 cm square of AlloMax will be harvested from the first 20 patients for histologic examination to determine wether or not there is neovascularization and collagen deposition.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Allomax: The cohort consists of immediate breast reconstruction patients who have AlloMax placed at the time of their tissue expander based immediate breast reconstruction.

SUMMARY:
The study is a prospective multi-centered cohort study designed to determine the safety and efficacy of AlloMax in immediate expander-based breast reconstruction. Specifically, the study is designed to determine if sterility of human acellular dermal matrix results in a lower incidence of infection and seroma. The study will determine if gamma radiation, as a method of terminally sterilizing human acellular dermal matrix, has a negative impact on graft incorporation into the host tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients having immediate breast reconstruction with tissue expanders
* Unilateral or bilateral reconstructions
* Ages 25 - 65
* All breast cancer stages and types

Exclusion Criteria:

* BMI > 35
* Active smokers
* Diabetics
* History of radiation or planned radiation
* Immunocompromised patients

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who opt for immediate breast reconstruction with tissue expanders from clinic.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Plastic Surgery, McLean, Virginia, United States

REFERENCES:
- [Derived] Venturi ML, Mesbahi AN, Boehmler JH 4th, Marrogi AJ. Evaluating sterile human acellular dermal matrix in immediate expander-based breast reconstruction: a multicenter, prospective, cohort study. Plast Reconstr Surg. 2013 Jan;131(1):9e-18e. doi: 10.1097/PRS.0b013e3182729d4f. PMID 22990174